CLINICAL TRIAL: NCT05990296
Title: Evaluating Strategies to Improve Guideline Directed Medical Therapy: The GDMT Research, Education & Assist Trial for Heart Failure Care (GREAT-HF Care)
Brief Title: Evaluating Strategies to Improve Guideline Directed Medical Therapy: The GDMT Research, Education & Assist Trial for Heart Failure Care
Acronym: GREAT-HF Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Stephen Voyce, Associate Professor, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-1031
Record Dates: First submitted 2023-07-31; First posted 2023-08-14 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction
Keywords: Heart Failure with Reduced Ejection Fraction; Guideline Directed Medical Therapy; Angiotensin-neprilysin inhibitors (ARNI); Sodium-glucose cotransporter 2 inhibitors (SGLT2i); Clinical Decision Support; Best Practice Alert; Pharmacist; Education; Behavioral Economics; Best Practice Advisory
MeSH Terms: conditions — Heart Failure | interventions — Caffeine; Educational Status; Drug Interactions

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized (at clinician level) design in terms of assignment to no-intervention control, multiprong CDS with GDMT order set, and multiprong CDS with referral to pharmacist co-management, and non-randomized (at clinic level) in terms of assignment to education versus delayed education arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control (No Intervention): Clinicians in this arm will not receive CDS or focused education and will experience usual care.
- Multiprong CDS with GDMT order set (Experimental): Clinicians and patients with HFrEF in this arm will receive electronic notification of GDMT care gaps encouraging treatment options. The CDS will inform, encourage, and facilitate prescribing of GDMT via a focused order set.
  Interventions: Behavioral: Multiprong CDS with GDMT order set
- Multiprong CDS with referral to pharmacist co-management (Experimental): Clinicians and patients with HFrEF in this arm will receive electronic notification of GDMT care gaps encouraging treatment options. The clinician-facing BPA will include an option to refer patients to embedded pharmacist co-management. Pharmacists are expected to meet with patients and optimize GDMT through a collaborative practice agreement with clinicians.
  Interventions: Behavioral: Multiprong CDS with referral to pharmacist co-management
- Focused education (Experimental): Clinicians in this arm will receive focused education and no CDS.
  Interventions: Behavioral: Focused education
- Multiprong CDS with GDMT order set + focused education (Experimental): Clinicians in this arm will receive focused education in addition to clinician BPA heads-up and BPA with GDMT order set for their eligible patients with HFrEF.
  Interventions: Behavioral: Multiprong CDS with GDMT order set; Behavioral: Focused education
- Multiprong CDS with referral to pharmacist co-management + focused education (Experimental): Clinicians in this arm will receive focused education along with clinicians/patient CDS. The clinician-facing BPA will include an option to refer patients to embedded pharmacist co-management. Pharmacists are expected to meet with patients and optimize GDMT through a collaborative practice agreement with clinicians.
  Interventions: Behavioral: Multiprong CDS with referral to pharmacist co-management; Behavioral: Focused education

INTERVENTIONS:
Behavioral: Multiprong CDS with referral to pharmacist co-management — Accepting the clinician-facing BPA default recommendation will have eligible patients within this arm referred to embedded pharmacist co-management. Pharmacists are expected to meet with patients and optimize GDMT through a collaborative practice agreement with clinicians. Clinicians will also be exposed to an interruptive advisory upon chart entry as a notification to physicians on GDMT consideration. Patient responses to a pre-visit questionnaire encouraging them to ask about better treatment options will also be shown to clinicians within the interruptive BPA if completed in advance by the patient.
  Other Names: Opt-out default; Active choice; Advisory; Alert
  Arms: Multiprong CDS with referral to pharmacist co-management; Multiprong CDS with referral to pharmacist co-management + focused education
Behavioral: Multiprong CDS with GDMT order set — Accepting the clinician-facing BPA default recommendation will open an order set for GDMT that lists common recommended options in such a way that facilitates optimal prescribing. Clinicians will also be exposed to an interruptive advisory upon chart entry as a notification to physicians on GDMT consideration. Patient responses to a pre-visit questionnaire encouraging them to ask about better treatment options will also be shown to clinicians within the interruptive BPA if completed in advance by the patient.
  Other Names: Opt-out default; Active choice; Default order of options; Advisory; Alert
  Arms: Multiprong CDS with GDMT order set; Multiprong CDS with GDMT order set + focused education
Behavioral: Focused education — A series of focused, interactive education sessions will train clinicians in why, when, and how to prescribe GDMT to patients, with incentives such as continuing medical education (CME) credits, and with virtual and recorded options available to those who are unable to attend in-person meetings.
  Other Names: Education; Training; Interactive
  Arms: Focused education; Multiprong CDS with GDMT order set + focused education; Multiprong CDS with referral to pharmacist co-management + focused education

SUMMARY:
Heart failure with reduced ejection fraction (HFrEF) is associated with high mortality and adverse events (hospitalization or urgent outpatient visits for HF), along with diminished quality of life. Despite convincing data that evidenced-based, guideline-directed medical therapies (GDMT) improve mortality and heart failure-related events, there remains insufficient utilization of these life-saving drugs (evidence-based beta-blockers (EBBB), angiotensin-neprilysin inhibitors (ARNI)/ angiotensin converting enzyme inhibitors (ACEi)/ angiotensin receptor blockers (ARB), mineralocorticoid receptor antagonists (MRA) and sodium-glucose cotransporter 2 inhibitors (SGLT2i) in patients with HFrEF. The primary objective of this study is to implement and evaluate a multifaceted, interdisciplinary intervention to improve GDMT use, reduce mortality, and reduce future heart failure events in patients with HFrEF.

DETAILED DESCRIPTION:
This is a cluster randomized study designed to evaluate the effectiveness of interventions aimed at improving GDMT in patients with HFrEF. Clinicians stratified based on practice specialty, location, and pharmacist referral habits will be permuted block randomized to achieve 45%/45%/10% proportional distribution across the following arms respectively: (1) usual care, (2) multi-pronged clinical decision support (CDS) inclusive of a patient portal message about GDMT, an interruptive advisory upon chart entry as a notification to clinicians on GDMT consideration and a Best Practice Advisory (BPA) that includes a GDMT order set, and (3) multi-pronged CDS as in #2 but replacement of GDMT order set with referral to integrated clinical pharmacist co-management. Secondarily, each of the 5 clinical practice sites of roughly equal HFrEF patient loads were assigned to receive either an early or delayed education rollout. Exploratory analyses will look to determine the independent and incremental benefits of education with other interventional approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older AND
* Completed visit at included Geisinger cardiology outpatient clinics (office visit or telemedicine) AND
* Clinicians are on a list of currently active Geisinger clinicians in outpatient cardiology clinics who can prescribe heart failure medications AND
* Active problem list diagnosis of HFrEF at time of Cardiology clinic encounter OR Left Ventricular Ejection Fraction (LVEF) < 40: most recent to the cardiology clinic encounter within 2 years of the visit.

Exclusion Criteria:

* Currently in hospice or palliative care (ICD 10 code: Z51.5)
* Patient is allergic to each category of GDMT
* Patient is prescribed medications from all four categories of GDMT, including ARNI specifically

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4306 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-05-17 (Actual)

PRIMARY OUTCOMES:
HF GDMT prescription increased (yes/no) | Within 30 days of index visit
  New GDMT HF medication class added, switch to ARNI from ACE/ARB, or upward dose titration of existing GDMT HF medication.

SECONDARY OUTCOMES:
HF GDMT prescription increased (yes/no) | Within 60 and 90 days of index visit
  New GDMT HF medication class added, switch to ARNI from ACEi/ARB, or upward dose titration of existing GDMT HF medication.
Addition of SGLT2i or ARNI for HFrEF (yes/no) | Within 30, 60 and 90 days of index visit
  New prescriptions for SGLT2i and/or ARNI or switch from ACEi/ARB to ARNI

OTHER OUTCOMES:
All-cause mortality, emergency visit for heart failure or hospitalization for heart failure | Within 365 days of index visit
  Patient death (yes/no), patient with emergency visit with a primary diagnosis of heart failure (yes/no) or admitted for inpatient hospitalization with primary diagnosis of heart failure (yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- Geisinger Cardiology Clinics, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT05990296/Prot_SAP_000.pdf